CLINICAL TRIAL: NCT01563939
Title: Patient-controlled Intravenous Analgesia With Remifentanil Infusion for Labour: is Demand Bolus Required for Optimal Analgesia
Brief Title: Patient-controlled Intravenous Analgesia With Remifentanil Infusion for Labour
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment.
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-02
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Labour analgesia; Pregnancy; IVPCA
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous infusion (Active Comparator): Remifentanil administered by continuous IV infusion, with stepwise increase in infusion rates and placebo demand bolus of normal saline.
  Interventions: Drug: Remifentanil
- Demand Bolus (Active Comparator): Demand bolus of remifentanil with stepwise increase in bolus dose and placebo continuous infusion of normal saline.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Remifentanil IV for continuous infusion: 0.025mcg/kg/min, increased by 0.025mcg/kg/min every 15 min if patient is not satisfied, to a maximum of 0.15mcg/kg/min.
  Remifentanil IV for demand bolus: 0.2 mcg/kg, lockout 2 min, incrementally increased if patient is not satisfied by 0.2 mcg/kg to a maximum of 1.2 mcg/kg.
  Other Names: remifentanil hydrochloride

SUMMARY:
Epidural analgesia for pain relief in labor may not be suitable for all patients, and intravenous patient controlled analgesia (IV PCA) with opioids offers the best alternative. The purpose of this study is to assess the effectiveness of two methods remifentanil administration in the form of either an infusion or PCA demand bolus (intravenous injection of a single dose over a short period of time). Currently, our hospital gives remifentanil by demand bolus, however it may be equally effective, with less side effects, to give the drug as an infusion.

DETAILED DESCRIPTION:
The study will be conducted as a randomized trial with two arms: Group I- continuous infusion of remifentanil with stepwise increase in infusion rates and Group II- demand bolus only with stepwise increase in bolus dose, as per the patient's analgesic requirement. Visual analog scores will be the primary outcome. Maternal and fetal side effects will be recorded. The results of this study will determine the regimen that suits the patients needs for painless labor with high efficacy, less adverse effects and a higher patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Term pregnancy in labour with singleton fetus in cephalic presentation
* Patients requesting systemic analgesia
* Patients with contraindication for regional anesthesia without fetal compromise (coagulopathy, thrombocytopenia, refusal, etc.)

Exclusion Criteria:

* Refusal to sign written informed consent
* Inability to communicate in English
* Opioid dependence or addiction
* Patients on Methadone
* Allergy or hypersensitivity to remifentanil
* Fetal heart rate abnormalities
* Fetal congenital anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours
  Verbal Numeric Rating Scale (VNRS) from 0 to 10 (where 0 = no pain and 10 = worst pain felt), approximately every hour, throughout labour.

SECONDARY OUTCOMES:
Maternal satisfaction | 24 hours
  Maternal satisfaction rated from 0-10, throughout labour
Consumption of remifentanil | 24 hours
  remifentanil consumed in mg/hr
Crossover to epidural | 24 hours
  Time to crossover if the patient decides to have an epidural
Side effects | 24 hours
  Sedation score, Heart Rate, Blood Pressure, Nausea, Vomiting, Pruritis
Fetal & Neonatal outcomes | 48 hours
  Non-reassuring fetal heart rate as determined by obstetrician, Neonatal weight, Apgar scores, naloxone administration, need for resuscitation, NICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada